CLINICAL TRIAL: NCT04031586
Title: The Role of a Nutritional Program on Delivery of Nutritional Services and Cost of Care in Children With Cancer in Nicaragua
Brief Title: Delivery of Nutritional Services in Nicaragua
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR7379
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Nutrition in Cancer Survival and Treatment
Keywords: Malnutrition; Childhood Cancer; Central America; Nicaragua
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children diagnosed with Solid Tumors: Children diagnosed with solid tumors in Managua, Nicaragua in Central America

SUMMARY:
This study investigates nutritional status, at predefined points in therapy, and the association with outcomes in children and adolescents undergoing treatment for cancer in institutions under Asociación de Hemato-Oncología Pediátrica de Centro América (AHOPCA) consortium in Central America. The aim of the study is to examine the effects of the newly-established nutritional program aimed at improving the delivery of nutritional care and outcomes in children undergoing treatment for cancer in Central America.

DETAILED DESCRIPTION:
In low and middle-income countries, children with cancer are simultaneously dealing with malnutrition in high proportions. Without proper access to care and a minimal or basic level of care, these children are exposed to worse conditions. Studies have shown that more than half of the children with cancer are also malnourished at diagnosis. This increases children's risk of complications associated with the treatment as well as the abandonment of care, as well as decrease the level of survival rates. With an established nutritional education and clinical intervention program, the outcomes of these children can be improved, especially in Central America where the cancer rates and malnutrition is high, as shown by several studies.

ELIGIBILITY:
Inclusion Criteria:

* Recent diagnosis of childhood cancer (Solid Tumors)
* Recruited at diagnosis
* Under the age of 18 years

Exclusion Criteria:

* Other cancer diagnosis
* Palliative care patients

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with solid tumors in Children's Hospital Manuel de Jesus Rivera (CHMJR) in Nicaragua will be recruited at diagnosis. A total of 300 patients are anticipated for the study in AHOPCA affiliated institution. Patients will be recruited and consented (including parents) by a designated researcher. Demographics is collected from medical records, and other required data will be collected from charts and/or assessed by the designated researcher or clinician. Accrual is anticipated to take place over a 3-year period. All data collection will occur on routine clinical visits or during hospitalization, as per treatment protocol, not requiring otherwise unscheduled visits to the hospital. Determination of time-points coincides with variations in therapy as per the treatment protocols followed by the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of malnutrition | Up to 3 years
  Determine the change in malnutrition by comparing nutritional status measured by anthropometric data at diagnosis and during and end of treatment.
Rate of utilization of nutritional interventions | Up to 3 years
  Impact on the delivery of nutritional services, defined as utilization of nutritional interventions. Information on utilization of nutritional services will be collected on a medical nutrition support (MNS) case report form, which collects information on the provision of enteral feeds (nasogastric feeds, gastrostomy feeds), oral nutrition supplements (e.g. Pediasure®, Ensure®) and days of total parenteral nutrition (TPN) over the previous phase of treatment. The MNS form also provides information on the brand of nutritional formula and the prescribed dose (i.e. amount in grams of supplement per day). If enteral feeds are administered, the formula, rate, and duration are reported. The responses collected on the MNS form will be used to determine the rate of utilization of nutritional interventions.

SECONDARY OUTCOMES:
Cumulative number of grade 3/4 toxicities | Up to 3 years
  Investigate association of nutritional status and the occurrence of grade 3/4 toxicities using NCI Common Toxicity Criteria (CTC).
Survival rate | Up to 3 years
  Survival is defined by both overall survival (time from enrollment to death from any cause) and event-free survival (time from enrollment to the first episode of relapse, disease progression or death).
Disease relapse rate | Up to 3 years
  Investigate the association of nutritional status and disease relapse
Rate of chemotherapy dose reductions | Up to 3 years
  The rate of chemotherapy dose reductions will be measured.
Number of treatment delays (in days) | Up to 3 years
  The number of treatment delays will be measured in days
Total duration of hospital stay | Up to 3 years
  The total duration of hospital stay will be measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Ladas, Phd, RD, Principal Investigator — Columbia University; Roberta Ortiz, MD, Principal Investigator — Children's Hospital Manuel de Jesus Rivera (CHMJR)
Locations (1):
- Children's Hospital Manuel de Jesus Rivera (CHMJR), Managua, Nicaragua

IPD SHARING:
Plan to Share IPD: No